CLINICAL TRIAL: NCT01804231
Title: A Prospective Study of Hybrid PET/MRI in the Evaluation of Men With Suspected Prostate Cancer Recurrence Following Definitive Local Therapy
Brief Title: Prospective Study Using Hybrid PET/MRI to Evaluate Men With Suspected Recurrence Following Treatment for Prostate Cancer
Acronym: IGPC-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IGPC-3; CTP-87515 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PET; MRI; Hybrid; Recurrence; Fluorocholine
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FCH PET/MRI imaging (Other): Patients eligible for the study will have an 18F-FCH PET/MRI in addition to standard of care clinical assessment and imaging (CT and bone scan)
  Interventions: Other: 18F-FCH PET/MRI imaging

INTERVENTIONS:
Other: 18F-FCH PET/MRI imaging — Patients will first undergo screening to ensure eligibility. If eligible, they will undergo one scan in a Hybrid PET/MRI scanner using 18F-FCH as the radiolabeled tracer.

SUMMARY:
Evaluate the impact of hybrid 18F-Fluoro-choline (18F-FCH) PET/MRI imaging on the clinical management of men with suspected recurrent prostate cancer post prostatectomy or radiotherapy.

We hypothesize that hybrid imaging incorporating 18F-FCH PET/MRI imaging will be feasible and will lead to changes in management decisions among men being re-staged for suspected prostate cancer recurrence post-surgery or radiation who are potentially eligible for local salvage therapy.

DETAILED DESCRIPTION:
The study will be a non-randomized, prospective study of men with suspected local recurrence of prostate cancer post-prostatectomy or radiation with negative bone and CT scans. Hybrid PET/MRI using 18F-FCH will be obtained and a consensus staging report generated for the attending clinician. Clinical management questionnaires completed by the study investigator will be obtained pre and post imaging in order to gauge the impact of the hybrid imaging on clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer with rising prostate specific antigen (PSA) post prostatectomy or radiotherapy
* Suspected recurrence based on PSA rise measured on 3 occasions at least 3 months apart and an absolute PSA > 0.2 ng/mL
* Bone scan and CT scan of the abdomen and pelvis negative for metastatic disease

Exclusion Criteria:

* Evidence of metastatic disease
* Contradiction to 18F-FCH PET scan
* Contraindication to MRI

Ages: 19 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Frequency in change of clinical management based on results of 18F-FCH PET/MRI | Within 2 weeks of study scan
  A questionnaire to assess the planned management will be completed by the investigator before and after provision of the results of the 18F-FCH PET/MRI to determine if the information provided by 18F-FCH PET/MRI influences the preferred plan of management

SECONDARY OUTCOMES:
Number of lesions identified with 18F-FCH based on consensus reporting | Within 2 weeks of study scan

OTHER OUTCOMES:
Concordance between MRI and 18F-FCH PET for lesion identification | Within 2 weeks of study scan
  Lesions identified on the 18F-FCH MRI/PET will be examined to determine what proportion of lesions are present on both MRI and PET imaging versus what proportion of lesions are present on only one of MRI or PET

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Glenn S Bauman, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada